CLINICAL TRIAL: NCT00523679
Title: SMART (Symbicort Maintenance And Reliever Therapy): Reassure Program for Patients Using Symbicort Turbuhaler as Maintenance and Reliever Therapy in Korean Clinical Practice
Brief Title: Symbicort SMART (Symbicort Maintenance And Reliever Therapy)
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-RKR-SYM-2007/1
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: Asthma; Symbicort; SMART; inhaler; compliance; Naturalistic; Observational
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the extent of Symbicort use in patients prescribed Symbicort as maintenance and reliever therapy.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients prescribed Symbicort as maintenance and reliever therapy, according to the label, before inclusion in this program.

Exclusion Criteria:

* Since this programme intends to describe Symbicort use in routine clinical practice when prescribed as Symbicort maintenance and reliever therapy, there are no programme specific exclusion criteria, other than: involvement in the planning and conduct of the programme (applies to both AstraZeneca staff or staff at the investigational site)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital Outpatient Clinics
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-07; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Woo Bahn, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Seoul, Jongro-gu
  - Research Site, Seoul, Kangnam-gu
  - Research Site, Seoul, Songpa-gu